CLINICAL TRIAL: NCT01294566
Title: A Randomized, Placebo Controlled Dose Escalation Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Oral Doses of GSK1322888 in Healthy Caucasian and Japanese Asian Adult Subjects
Brief Title: FTIH to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Oral Doses of GSK1322888 in Healthy Caucasian and Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 114422
Record Dates: First submitted 2011-02-03; First posted 2011-02-11 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Gastroparesis
Keywords: safety; motilin agonist; single dose; ascending dose; GSK1322888; migrating motor complex; tolerability; FTIH; gastric emptying
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): GSK1322888 (1 mg, 2 mg, 5 mg, 10 mg; 6 subjects) and Placebo (32 subjects)
  Interventions: Drug: GSK1322888; Drug: Placebo
- Cohort 2 (Experimental): GSK1322888 (20 mg, 40 mg, 80 mg, and dose to be determined; 6 subjects) and Placebot (2 subjects)
  Interventions: Drug: GSK1322888; Drug: Placebo

INTERVENTIONS:
Drug: GSK1322888 — 1 mg, 5 mg or 25 mg capsule
Drug: Placebo — matching placebo capsules

SUMMARY:
This study is the First Time In Human study for the motilin receptor agonist, GSK1322888. GSK1322888 is a potent and selective small molecule motilin receptor agonist, distinct from the motilide compound structures. The aims of this study are to assess the safety, tolerance, and pharmacokinetics of single oral doses of GSK1322888 and to identify a well-tolerated and safe dose that will accelerate gastric emptying of a 13C stable isotope-labeled test meal in healthy volunteers.

The study will include assessment of ECGs, vital signs, safety laboratory sampling, adverse events, pharmacokinetics, and the 13C-Octanoic Acid Breath Test to measure gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin < or =1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician
* Male or female between 18 (20 for Japanese) and 65 years of age inclusive
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods
* Body weight > or = 50 kg and BMI within the range 18.5 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent
* Average QTc, QTcB or QTcF < 430 msec.
* For Japanese subjects Japanese ancestry defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese.

Exclusion Criteria:

* Hepatitis B or Hepatitis C positive
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* HIV positive
* History of regular alcohol consumption within 6 months of the study
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) prior to the first dose of study medication
* History of sensitivity to any of the study medications, or components thereof
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Subjects will be screened such that those subjects exhibiting rapid gastric emptying rates (t½b < 75 min) will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11-29 (Actual); Primary Completion 2011-03-23 (Actual); Study Completion 2011-03-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events following single oral doses of GSK1322888 | 1 week post dose
  includes abnormal clincal lab values, ECGs, vital signs
pharmacokinetics of GSK1322888 following single, oral doses | 48 h post dose
  includes AUC, Cmax, tmax, and t1/2

SECONDARY OUTCOMES:
gastric emptying of a radio-labeled test meal, as measured by the 13C-octanoic acid breath test following single oral doses of GSK1322888 | 4 h
  includes gastric half emptying time, gastric emptying coefficient
dose/exposure response relationship for gastric emptying of a radio-labeled test meal, as measured by the 13C-octanoic acid breath test following single oral doses of GSK1322888 | 48 h
  dose response of GSK1322888 on gastric emptying
dose proportionality following single dose administration | 48 h
steady-state PK based on single dose data | 28 h
accumulation based on single dose data | 48 h
ethnicity differences in safety, tolerability, pharmacokinetics, and pharmacodynamics between volunteers of Caucasian or Japanese ethnicity | 1 week
  difference in adverse events between ethnicities

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114422 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114422?search=study&search_terms=114422#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114422 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register